CLINICAL TRIAL: NCT01052207
Title: Prevalence of Oxidative Stress in Critically Ill Children and Its Relationship to Adrenal Insufficiency; a Pilot Study
Brief Title: Pilot Study Assessing Oxidative Stress in Children
Acronym: OxStress
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Kiran Hebbar, Assistant Professor, Emory University
Other Study IDs: IRB00034236
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-05

CONDITIONS: Adrenal Insufficiency; Critical Illness
Keywords: Biological Response Modifiers; Endocrinology; Hormone Dysfunction; Hormones; Neuroendocrinology
MeSH Terms: conditions — Adrenal Insufficiency; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum from critically ill patients
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Critically Ill Patients: Evaluation of Oxidative Stress, Glucocorticoid Receptor function, and Adrenal Insufficiency amongst critically ill pediatric patients. Serum, and when available endotracheal samples, will be obtained within 24 hours of admission and at 5 days provided patients are 1) still in the PICU and 2) blood draws and endotracheal aspirates are part of their standard of care. Endotracheal aspirates will be sent on day 14, 21, and 28 provided patients are intubated and require suctioning as part of their standard of care.
- Healthy Controls: Healthy controls will be evaluated and defined as those who do not have any chronic medical condition, are not on steroids (inhaled or oral), and have not received steroids or etomidate in the last month. Given the time and need for multiple lab draws low dose adrenocorticotropin (ACTH) testing will not be done in healthy patients, nor will tracheal aspirate samples be obtained.

SUMMARY:
Role fo oxidative stress in adrenal insufficiency has not been studied. The degree of oxidative stress and it's role in pediatric critical illness is unknown. Potential for significant alterations to many of thew body's regulatory pathways may result from severe oxidative stress. Further is needed to delineate what if any role oxidative stress may play

DETAILED DESCRIPTION:
Adrenal insufficiency (AI) is common in critically ill children and adults. AI is a condition in which the adrenal glands, located above the kidneys, do not make enough hormones or our body is unable to use the hormones made. A hormone is a chemical that helps control different kinds of body functions. The hormones being studied can influence blood pressure and how fast the heart beats. Doctors want to know why children need extra hormones when they are critically ill. In our pediatric intensive care unit (PICU) we treat AI with a set of standard orders. By doing this, we have shown that AI is common in many types of sickness and that blood pressure improves when extra hormones are given. We also found that people's heart and blood pressure did not always match the level of a certain hormone, called cortisol, in their blood.

Since cortisol levels alone don't always show AI, and children with normal hormone levels still benefit from steroids, doctors are looking for a better understanding of AI. Finding reasons that children develop AI may help doctors find other ways to improve AI.

One promising focus of AI is the role of oxidative stress (OS). OS is a term used to describe a group of chemical reactions that involve oxygen. Emory's adult intensive care units have shown a significant increase in OS in critically ill patients. Normally our body's cortisol acts by binding to glucocorticoid (a class of hormone) receptors (GR) within cells. Many studies have shown that OS increases steroid resistance by changing the GR structure and function. Studies involving OS and GR problems have not been done with children.

We aim to:

1. Find out how many sick children have OS in the PICU.
2. Find out the normal OS level of healthy children.
3. Decide if OS causes adrenal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

Critically Ill subjects:

1. All patients, birth-18 years, admitted to the pediatric intensive care unit that require blood to be drawn as part of medical management consistent with "standard of care".
2. Admission to the PICU within the last 24 hours.
3. Subjects' legal guardian shall possess the ability to understand the purposes and risks of the study and provide an informed consent signature.

Healthy control subjects:

1. All healthy children, birth-18 years, who are having semi-elective magnetic resonance imaging (MRI) that require peripheral intravenous (PIV) catheters placed to provide sedation.

Exclusion Criteria:

Critically Ill subjects:

1. Have received steroids within the last 30 days.
2. Pre-existing/known neuroendocrine disorder, including but not limited to disorders of the hypothalamus, pituitary, adrenal, pancreas, or thyroid gland.
3. Have been treated at anytime with antipsychotic medication.
4. Human immunodeficiency virus (HIV) positive.
5. Patients who have received etomidate.
6. Patients weighing less than or equal to 6 kilograms.
7. Developmentally delayed.
8. Medical urgency preventing timely administration of the consenting process, or any condition that, in the opinion of the attending physician, would place the patient at undue risk by participating.
9. Other technical considerations that would prevent the timely acquisition of sufficient samples such as (but not limited to) hour of admission or absence of a study team member.
10. Parent or legal guardian (or patient when applicable) refuses to sign informed consent.

Healthy control subjects:

1. Have received steroids within the last 30 days.
2. Have a pre-existing/known neuroendocrine disorder, including but not limited to disorders of the hypothalamus, pituitary, adrenal, pancreas, or thyroid gland.
3. Have been treated at anytime with antipsychotic medication.
4. Human immunodeficiency virus (HIV) positive.
5. Patients who have received etomidate.
6. Patients weighing less than or equal to 6 kilograms.
7. Developmentally delayed.
8. Medical urgency preventing timely administration of the consenting process, or any condition that, in the opinion of the attending physician, would place the patient at undue risk by participating.
9. Other technical considerations that would prevent the timely acquisition of sufficient samples such as (but not limited to) hour of admission or absence of a study team member.
10. Parent or legal guardian (or patient when applicable) refuses to sign informed consent.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Population 1 consists of critically ill patients being care for in quaternary PICU.
  Population 2 consists of relatively healthy children undergoing MRI for sedation
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Hebbar, MD, FCCM, Principal Investigator — Emory University & Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Critically Ill Patients: Evaluation of Oxidative Stress, Glucocorticoid Receptor function, and Adrenal Insufficiency amongst critically ill pediatric patients. Serum, and when available endotracheal samples, will be obtained within 24 hours of admission and at 5 days provided patients are 1) still in the PICU and 2) blood draws and endotracheal aspirates are part of their standard of care. Endotracheal aspirates will be sent on day 14, 21, and 28 provided patients are intubated and require suctioning as part of their standard of care.
  Cortrosyn: Subjects : a 1 microgram (mcg) dose of Cosyntropin via intravenous access. After 30 minutes, blood samples collected.
Period: Overall Study
Arm/Group | Critically Ill Patients | Healthy Controls
Started | 60 | 42
Completed | 60 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Critically Ill Patients | Healthy Controls | Total
Number analyzed (Participants) | 60 | 42 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (5.6) | 8 (4.5) | 9.7 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 36 | 19 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 15 | 54
  White | 16 | 23 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 57 | 40 | 97
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 42 | 102

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Logistic Organ Dysfunction Score in Critically Ill Children
Description: Pediatric Logistic Organ Dysfunction also known as the PELOD Score is a marker of severity of illness for Critically ill children. The PELOD includes six organ dysfunctions and 12 variables.
  To calculate the PELOD score, each organ dysfunction received points for the single variable associated with the most points. The minimum number that can be assigned to an organ is 0 and the maximum number of points for an organ is 20, and the maximum possible PELOD score is 71. Organ dysfunction is identified if the score for any organ system was more than 0.
Time Frame: 1 years
Population: PELOD scores are not calculated for healthy controls. The score was developed to assess critically ill patients only.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Critically Ill Patients | Healthy Controls
Number analyzed (Participants) | 60 | 0
scores on a scale | 15.9 (13.7) |

2. Secondary Outcome: Establish the OS Profile of Healthy Children to Act as Controls and Help Establish the Normal Pediatric Baseline.
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Analysis of Clinical Data to Determine Correlation of OS With AI and Evaluation of OS as a Potential Biomarker.
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Observational blood draw study. Patient were not subjected to any risks
Description: this study did not place any patients at risk for harm. blood samples were only collected when routine blood (as part of patient care) was being drawn from an established centtral line or arterial line.
Groups:
- Critically Ill Patients: Evaluation of Oxidative Stress, Glucocorticoid Receptor function, and Adrenal Insufficiency amongst critically ill pediatric patients. Serum, and when available endotracheal samples, will be obtained within 24 hours of admission and at 5 days provided patients are 1) still in the PICU and 2) blood draws and endotracheal aspirates are part of their standard of care. Endotracheal aspirates will be sent on day 14, 21, and 28 provided patients are intubated and require suctioning as part of their standard of care.
  Cortrosyn: Subjects : a 1 microgram (mcg) dose of Cosyntropin via intravenous access. After 30 minutes, blood samples collected. only if deemed part of their clinical care
Arm/Group | Critically Ill Patients | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Critically Ill Patients (N=0) | Healthy Controls (N=0)
0 (Infections and infestations) | 0 | 0 — 0" Total Number of Participants at Risk This was not an intervention study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No